CLINICAL TRIAL: NCT00763256
Title: The Effect of Periodontal Treatment and the Use of Dentifrice on Glycaemic Control in Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004000841/2004/201
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases | interventions — Triclosan; Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Triclosan, Fluoride
- B (Placebo Comparator)
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Triclosan, Fluoride — subjects brushed their teeth twice daily with the study toothpaste for the assigned treatment period.
  Other Names: triclosan/fluoride/copolymer toothpaste
  Arms: A
Drug: Fluoride — subjects brushed their teeth twice daily with the study toothpaste for the assigned study treatment period.
  Other Names: current marketed fluoride only toothpaste
  Arms: B

SUMMARY:
To test effectiveness of dentifrice in maintaining periodontal health.

ELIGIBILITY:
Inclusion Criteria:

* Poor glycaemic control as evidenced by an HbA1c of >6.0% for the past 12 months
* Aged 18 to 75 years
* Able to give informed consent
* Minimum of 12 teeth
* Chronic periodontitis as indicated by periodontal probing depths >5mm on at least 6 teeth

Exclusion Criteria:

* Pregnancy
* Gross dental caries
* Prosthetic heart valves, a history of infective endocarditis or any other condition requiring antibiotic cover for dental treatment (rheumatic fever, mitral valve prolapse with regurgitation)
* Anticoagulant therapy (excluding asprin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Seymour, BDS, Principal Investigator — University of Otago
Locations (1):
- Logan Hospital Oral Health Clinic, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all subjects were recruited at the clinical site by the PI.
Pre-assignment Details: All subjects passed a medical exam and met the inclusion/exclusion criteria.
Groups:
- Active Comparator: triclosan/fluoride/copolymer toothpaste
- B - Placebo Comparator: fluoride only toothpaste
Period: Overall Study
Arm/Group | Active Comparator | B - Placebo Comparator
Started | 15 | 18
Completed | 8 | 8
Not Completed | 7 | 10
Not completed — Didn't return for appointments | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | B - Placebo Comparator | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (7.6) | 49 (11) | 51 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  Australia | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Levels in Blood
Description: Glycated hemoglobin (HbA1c) is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. In this study, blood is taken from each subject and HbA1c levels were measured at 12 months by Queensland Health Pathology Scientific Services (QHPSS).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Active Comparator | B - Placebo Comparator
Number analyzed (Participants) | 15 | 18
Percentage | 9.47 (2.2) | 10.27 (2.4)
Statistical Analysis 1: Comparison: Active Comparator vs B - Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

2. Primary Outcome: High Sensitivity CRP (C-Reactive Protein)
Description: CRP is a protein found in the blood and is a marker for inflammation in the body. Inflammation plays a role in the initiation and progression of cardiovascular disease. Blood is taken from each subject and CRP levels were measured at 12 months by Queensland Health Pathology Scientific Services (QHPSS).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Active Comparator | B - Placebo Comparator
Number analyzed (Participants) | 15 | 18
mg/L | 6.16 (5.5) | 5.37 (3.8)
Statistical Analysis 1: Comparison: Active Comparator vs B - Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

3. Primary Outcome: C-Peptide
Description: C-Peptide levels in blood indicate whether or not a person is producing insulin. This peptide is usually found in equal levels to insulin. C-peptide levels measured as a means of distinguishing type 1 diabetes and type 2 diabetes. Blood is taken from each subject and C-Peptide levels were measured at 12 months by Queensland Health Pathology Scientific Services (QHPSS).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Active Comparator | B - Placebo Comparator
Number analyzed (Participants) | 15 | 18
nmol/L | 1.20 (1.0) | 1.04 (0.6)
Statistical Analysis 1: Comparison: Active Comparator vs B - Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

4. Primary Outcome: Gingivitis Score (GI)
Description: Units on a scale 0 to 3 (0 = no inflammation,
  1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active Comparator | B - Placebo Comparator
Number analyzed (Participants) | 15 | 18
Units on a scale | 0.89 (0.2) | 0.88 (0.1)
Statistical Analysis 1: Comparison: Active Comparator vs B - Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

5. Primary Outcome: P. Gingivalis
Description: Subgingival plaque samples were collected from all interproximal (mesial) sites and pooled prior to assessment. The samples will be analysed for the presence of P. gingivalis, using real time PCR to quantitate the numbers of bacteria. P. gingivalis is a non-motile, gram negative, anaerobic, pathogenic bacteria. It is linked to periodontal disease and causes collagen degradation.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Pg/ng DNA
Arm/Group | Active Comparator | B - Placebo Comparator
Number analyzed (Participants) | 15 | 18
Pg/ng DNA | 209 [0 to 23688] | 22 [0 to 15982]
Statistical Analysis 1: Comparison: Active Comparator vs B - Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Active Comparator | B - Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less